CLINICAL TRIAL: NCT06990139
Title: Ventricular Tachycardia Ablation Through Radiation Therapy Consortium: Concept Description of an Observational Retrospective Multicentric Trial Via Matched Pair Analysis (VT-ARTr)
Brief Title: Ventricular Tachycardia Ablation Through Radiation Therapy Consortium: Concept Description of an Observational Retrospective Multicentric Trial
Acronym: VT-ART R
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CELLINI FRANCESCO, Clinical Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0001344/24
Record Dates: First submitted 2025-04-23; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: ventricular tachycardia; radioablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who have undergone SBRT: Within this group we find patients who have had all possible canonical treatments for the arrhythmia and also the stereotactic radiation treatment
- patients who have not undergone SBRT: Within this group we find patients who have had all possible canonical treatments for the arrhythmia, but not the stereotactic radiation treatment

SUMMARY:
Recurrent ventricular tachycardia (VT) is a potentially life-threatening arrhythmia in patients with structural heart disease. Despite the use of antiarrhythmic drugs, implantable cardioverter-defibrillators (ICDs), and radiofrequency catheter ablation, VT recurrence rates remain high-reaching up to 66% in some series. For patients with refractory VT who are not candidates for further ablation or surgical interventions, there is a significant unmet need for novel, effective, and non-invasive treatment options.

Stereotactic body radiation therapy (SBRT) has recently emerged as a promising approach for treating ventricular arrhythmias through a technique known as stereotactic arrhythmia radioablation (STAR). Preliminary studies, including a phase I/II clinical trial, have demonstrated a substantial reduction in VT burden-up to 99.9%-following treatment, with an acceptable safety profile. Reported adverse events have included manageable pericardial effusion, radiation-induced pericarditis, and pneumonitis. The growing body of evidence supports STAR as a feasible and effective alternative for selected patients with treatment-resistant VT.

The objective of this study is to evaluate the efficacy and safety of stereotactic radiotherapy as a non-invasive ablation technique for the treatment of ventricular tachycardia (VT) in patients with refractory arrhythmias in whom conventional therapies have failed.

This is a retrospective observational study aimed at comparing outcomes between patients who received stereotactic radioablation and those who did not. A matched-pair analysis will be used to adjust for baseline clinical characteristics and ensure comparability between groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory ventricular tachycardia (VT), as previously defined
* Age greater than 18 years
* Presence of an implantable cardioverter-defibrillator (ICD) for follow-up
* Not eligible for heart transplantation
* Estimated life expectancy of at least 1 year
* Ability to provide autonomous, informed consent to participate in the study

Exclusion Criteria:

* ICD interrogation demonstrating polymorphic VT
* Patients with INTERMACS class more than 4
* Patients with LVADs
* Patients with active neoplastic disease under oncological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at Fondazione Policlinico Gemelli IRCCS and in all centers that joined the protocol
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in VT episode frequency compared to the pretreatment period | Starting from three months before treatment until 3 months later
  The number of VT episodes during the 3 months prior to treatment will be compared to the number of episodes recorded during the 3-month period following the post-treatment blanking period. This comparison will help determine whether the treatment provides clinical benefits even at an early stage

SECONDARY OUTCOMES:
Change in antiarrhythmic drug burden compared to the baseline | 36 months
  The study aims to show whether radioablation treatment is associated with a significant reduction in the use of antiarrhythmic drugs compared to patients who did not undergo the procedure
Change in left ventricular end-diastolic volume compared to the baseline | 36 months
  Improvement in left ventricular end-diastolic volume, as assessed through specific tests performed by a cardiologist specializing in arrhythmology, especially the Echocardiogram, and a global electrophysiological evaluation
Change in left ventricular end-systolic volume compared to the baseline | 36 months
  Improvement in left ventricular end-systolic volume , as assessed through specific tests performed by a cardiologist specializing in arrhythmology , especially the Echocardiogram, and a global electrophysiological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Largo Francesco Vito 1, 00168, Rome (Italy), Rome, ROME, Italy

IPD SHARING:
Plan to Share IPD: Undecided